CLINICAL TRIAL: NCT00022919
Title: Analysis of Prostate Cancer Short-Term Cultures Utilizing Molecular Cytogenetic Methods
Brief Title: Analysis of Prostate Cancer Short-Term Cultures Using Molecular Cytogenetic Methods
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 010212; 01-HG-0212
Record Dates: First submitted 2001-08-16; First posted 2001-08-17 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-08

CONDITIONS: Prostate Cancer
Keywords: Microdissection; Chromosome; Karyotype; Tumor; Malignancy; Prostate Adenocarcinoma; Prostate Intraepithelial Neoplasia; Prostate Cancer; Prostate
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

SUMMARY:
This study will examine prostate tumor tissue cultures to try to identify genetic abnormalities that contribute to the cause or progression of the disease.

Patients with prostate cancer enrolled in the National Cancer Institute protocol 97-C-0147 (Collection of Serum and Tissue Samples from Patients with Biopsy-Proved or Suspected Malignant Disease) may be eligible for this study.

Specimens for tissue culture for this study will be obtained from tumors surgically removed from patients participating in NCI protocol 97-C-0146.

The findings of this study may lead to better methods of predicting the course of disease in individual patients.

DETAILED DESCRIPTION:
Prostate cancer is the most common solid tumor in American males and the most common malignancy among men in Western industrialized countries. Widespread testing for early detection of prostate cancer utilizing digital rectal examination and prostate specific antigen (PSA) has led to a significant clinical conundrum. Differentiating organ confined indolent disease from aggressive cancer has been imperfect. Nonetheless, increased detection has led to increased radical prostatectomies. A prevailing goal of the contemporary, ardent research seeks to discover a molecular biomarker for prognostication.

Given the limitations of the current knowledge of the molecular pathology of prostate cancer, there are several viewpoints regarding the process of tumorigenesis. However, a generally accepted hypothetical model describes normal prostatic epithelium progressing to a pre-malignant or low-grade prostatic intraepithelial neoplasia (PIN). Then, after further genetic alterations, a succession of histologically apparent adenocarcinoma--first confined, then metastatic, and finally refractory to hormone treatment ensues. Current molecular research has shown already complex genetics alterations at the high-grade prostatic intraepithelial neoplasia stage. Thus, invasive disease represents amplification or further aberration of precursor events. The seminal event or events have not been recognized and the undiscovered tumor suppressor gene or proto-oncogene may be a principal tumor marker.

The purpose of this study is to identify specific, shared, consistent, chromosomal rearrangements found in metaphase preparations for short-term cultures of pathologically identified and scored primary prostate tumors. These, tumor specimens will be obtained from patients enrolled in protocol (97-C-0147) by the NCI. Fresh tumor, taken from bi-valved specimens with one half undergoing tissue pathology, will be immediately placed in growth media and transferred as a coded specimen as a sample from patients selected and enrolled in protocol (97-C-0147). Informed consent will be obtained by participating investigators in the NCI protocol. The outcome measurement will be the characterization, or failure of characterization, of specific, shared consistent, chromosomal rearrangements. Current molecular cytogenetics technologies, primarily utilizing chromosomal microdissection, will be employed toward this goal. Ultimately, this research may help to focus further molecular studies towards the ultimate goal of finding a unique, cancer specific alteration.

ELIGIBILITY:
INCLUSION CRITERIA:

Only patients who have met pathologic criteria for prostate intraepithelial neoplasia or higher (determined by pathologists included in the NCI protocol) will be included for entry into this protocol.

EXCLUSION CRITERIA:

No prisoners, decisionally impaired, healthy volunteers, or lab personnel will be included in this study.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150
Dates: Start 2001-08; Study Completion 2004-08

CONTACTS AND LOCATIONS:
Locations (1):
- National Human Genome Research Institute (NHGRI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Reiter RE, Gu Z, Watabe T, Thomas G, Szigeti K, Davis E, Wahl M, Nisitani S, Yamashiro J, Le Beau MM, Loda M, Witte ON. Prostate stem cell antigen: a cell surface marker overexpressed in prostate cancer. Proc Natl Acad Sci U S A. 1998 Feb 17;95(4):1735-40. doi: 10.1073/pnas.95.4.1735. PMID 9465086
- [Background] Nupponen NN, Isola J, Visakorpi T. Mapping the amplification of EIF3S3 in breast and prostate cancer. Genes Chromosomes Cancer. 2000 Jun;28(2):203-10. PMID 10825005
- [Background] Nupponen NN, Visakorpi T. Molecular cytogenetics of prostate cancer. Microsc Res Tech. 2000 Dec 1;51(5):456-63. doi: 10.1002/1097-0029(20001201)51:53.0.CO;2-H. PMID 11074616